CLINICAL TRIAL: NCT06907940
Title: Upper Extremity Stability and Balance in Youth Basketball Players
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Star Balance Test Adolescent
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Balanced
Keywords: basketball

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amateur Basketball Football Team: Players of the Amateur Basketball Football Team will participate in our study, and after the demographic information of all participants is collected.

SUMMARY:
Ball games require extensive skill, including physical, technical, mental and tactical abilities. Among them, the physical abilities of the players show obvious effects on the players' own skills and the tactics of the team. It involves skillful moves that include shooting, defending, and dribbling. It requires repeated maximum effort, such as a.

DETAILED DESCRIPTION:
Endurance is defined as the strength of the physical and physiological characteristics of a basketball player to cope with fatigue. Flexibility is the ability of the athlete to use the range of motion he uses while demonstrating the movements, in every possible direction in the joint range.

ELIGIBILITY:
Inclusion Criteria:

* Being a basketball player
* Regular attendance at training sessions

Exclusion Criteria:

* Known neurological disorder
* Serious orthopedic disorders that prevent exercise
* cognitive impairment

Ages: 14 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: basketball player
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test | day 1
  Eight directions including anterior, superomedial, medial, inferomedial, posterior, inferolateral, lateral, and superolateral were marked on floor by tapes with scale and the angle between each strip of tape were 45°. The minimum unit of the UESEBT was 0.5 cm. Distances for analysis were normalized by dividing the right upper limb length of every participant, and then multiplying by 100.
Medicine Ball Throwing | day 1
  Individuals will be asked to take a position in front of a wall, with feet shoulder-width apart, to grasp the medicine ball with both hands. A medicine ball weighing three kg will be used in this test. Individuals will be asked to bring the medicine ball upside down and throw it forward.The distance the ball is thrown will be recorded
Upper extremity Y Test | day 1
  Upper extremity lengths are determined by measuring the distance between the C7 cervical vertebra processus spinosus and the middle fingertip of the athletes. In this position, the athletes are positioned perpendicular to the middle extension of the Y balance kit (the arm that makes an angle of 135° with the other ends). Afterwards, the athlete is asked to push the platform apparatus along the superior and inferior arms, which are lateral to the lateral side of his fixed hand, and take it to the last point it can take. Y balance scores were found using the reach distance and limb length in each direction.
Closed Kinetic Chain Upper Extremity Stability Test (TEST) | day 1
  Individuals were positioned in the push-up position, with their bodies aligned in a straight line when viewed from the side, with a distance of 90 cm between their hands. The athletes were asked to touch the dorsum of the dominant hand and the other hand within 15 seconds, and the total number of repetitions was recorded.
Push Up Test. | day 1
  The push-up test was performed with the participant pushing their arms off the floor until their elbows were straight while keeping their legs and back straight. This movement was repeated as many times as possible, ending when the subject stopped or the participant did not perform the push-ups properly or held the correct position several times.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu HR, Zhang YH, Mao Y, Ngo TL, Zhang Q, He G, Feng Z, Sun W, Wang XQ. Validity and reliability of upper extremity star excursion balance test in adolescent swimmers. J Exerc Sci Fit. 2023 Apr;21(2):210-217. doi: 10.1016/j.jesf.2023.02.003. Epub 2023 Feb 27. PMID 36923209